CLINICAL TRIAL: NCT05265403
Title: Evaluation of High-Performance, Customized, Rapidly-Manufacturable Prosthetic Feet That Provide Improved Mobility
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Massachusetts Institute of Technology (Other)
Collaborators: Hanger Clinic: Prosthetics & Orthotics (Other)
Responsible Party: Sponsor
Other Study IDs: 2106000399
Record Dates: First submitted 2022-01-26; First posted 2022-03-03 (Actual); Last update posted 2022-04-12 (Actual); Status verified 2022-02

CONDITIONS: Amputation of Lower Limb Below Knee
Keywords: transtibial amputation; below knee amputation; prosthetic device design; biomechanics

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Below knee amputees: Adult, unilateral trans-tibial amputees (amputation is below the knee and only on one side) who will wear and test our prototype prosthetic feet
  Interventions: Drug: Commercially-available energy storage and return prosthetic foot; Device: MIT-Lower Leg Trajectory Error (LLTE) customized prosthetic feet

INTERVENTIONS:
Drug: Commercially-available energy storage and return prosthetic foot — Each patient will walk in the Freedom Highlander, a commercially-available energy storage and return prosthetic foot. The foot will be sized based on the patient's foot size and weight.
  Other Names: Freedom Highlander
Device: MIT-Lower Leg Trajectory Error (LLTE) customized prosthetic feet — Each patient will walk in prosthetic feet designed by the researchers at MIT. These feet will be customized for the user based on their body size (ie, height, foot length) and weight.

SUMMARY:
The purpose of this research is to design a high-performance, customized, and rapidly- manufacturable passive prosthetic foot for use in the United States. We are currently testing an early stage prototype and would like user input before pursuing additional clinical testing. Participants will be asked about their current prosthesis type and use, amputation side and cause, and activity level. We will take measurements of height, weight, and length of the participant's residual limb. The participant will be asked to walk in several prosthetic foot conditions in multiple walking activities, and the visit should last approximately four hours.

For each prosthetic foot, a trained prosthetist will fit the foot (either a prototype foot or a commercially available K3/K4 foot) to the prosthesis. The patient will then walk around the room until they feel comfortable. They may initially walk using a gait belt or between parallel bars based on comfort level and an evaluation by the prosthetist. Once they feel comfortable walking on level ground at a normal speed and the prosthetist feels that they will be safe performing more challenging walking activities, the participant will perform different walking activities (such as walking on flat ground at different speeds, walking up/down ramps, and walking up/down stairs). They will then be asked to tell the investigator what they like and dislike about the prosthetic foot.

DETAILED DESCRIPTION:
The purpose of this research is to design a high-performance, customized, and rapidly- manufacturable passive prosthetic foot for use in the United States. We are currently testing an early stage prototype and would like your input before pursuing additional clinical testing. The Global Engineering and Research (GEAR) Laboratory at the Massachusetts Institute of Technology (MIT) has developed a novel design framework for creating high-performance, passive prosthetic feet. By incorporating commercial aesthetic and functional requirements, we hypothesize that we can use this design methodology to create high-performance prosthetic feet that can be customized and provided at scale in the United States.

Participants will be asked about their current prosthesis type and use, amputation side and cause, and activity level. We will take measurements of height, weight, and length of the participant's residual limb. The participant will be asked to walk in several prosthetic foot conditions in multiple walking activities, and the visit should last approximately four hours.

For each prosthetic foot, a trained prosthetist will fit the foot (either a prototype foot or a commercially available K3/K4 foot) to the prosthesis. The patient will then walk around the room until they feel comfortable. They may initially walk using a gait belt or between parallel bars based on comfort level and an evaluation by the prosthetist. Once they feel comfortable walking on level ground at a normal speed and the prosthetist feels that they will be safe performing more challenging walking activities, the participant will perform different walking activities (such as walking on flat ground at different speeds, walking up/down ramps, and walking up/down stairs). They will then be asked to tell the investigator what you like and dislike about the prosthetic foot.

Participants may also be asked to walk while wearing inertial measurement units (IMU's), which are wearable devices similar in size to a pedometer or wrist watch. These devices will record the acceleration of the limbs, which will allow us to understand how people walk in the different prosthetic feet. We will attach the IMU's using their elastic bands, and we will attach necessary wires with hypoallergenic tape. Wearing the IMU's, the participant will walk back and forth in the room while the sensors record information about how you are walking. They may rest at any time.

ELIGIBILITY:
Inclusion Criteria:

* Unilateral transtibial amputation
* Aged between 18-65 years
* Body mass index between 18.5-29.9 (healthy weight)
* Daily use of their clinically-prescribed prosthesis for ambulation without an assistive device
* Classified as at least a Medicare Functional Classification Level K3 (defined as a patient who is a typical unlimited community ambulator)
* Experience walking with a prosthesis for at least one year
* Residuum and amputated side in good condition (e.g., no adherent scars, lesions, ulcers, or infections)
* Normal or corrected vision
* Ability to walk continuously for 45 minutes without undue fatigue or health risks.

Exclusion Criteria:

* Subjects who weigh more than 200 pounds
* Poor fitting prosthetic socket
* Skin problems on the residual limb
* Co-morbidities or pathologies (other than the amputation) or medications that would affect the sound limb, spine, balance, or stability
* Decision by prosthetists at Hanger that walking on the prototype limb may pose higher than minimal risk for a potential subject.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects with a unilateral transtibial amputation will be recruited through the Hanger Clinic. Subjects will likely be recruited who live in the Salt Lake City, Utah area, where data will be collected. Potential subjects will be screened to ensure that they satisfy the inclusion criteria. Screening will take place during the recruitment process either in person at the clinic or when the subject makes contact with the investigator. Subjects will be asked questions to ensure they meet the study inclusion criteria.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2022-03-03 (Actual); Primary Completion 2022-07-30 (Estimated); Study Completion 2022-08-31 (Estimated)

PRIMARY OUTCOMES:
Number of patients who prefer each prosthetic foot tested for each walking activity | At the end of study completion, after ~4 hours of total time on a single day to acclimate to all prosthetic feet tested
  For each walking activity, subjects will qualitatively select which foot option they prefer for each activity (ie, standing, walking at varied speeds on level ground, and walking up/down ramps). Subjects will provide this information through a questionnaire where they indicate their preferred foot for each activity.
Mean difference in prosthetic foot evaluation score between prototype prosthetic feet and commercial prosthetic feet, as assessed by a self-reported questionnaire | At the end of study completion, after ~4 hours of total time on a single day to acclimate to all prosthetic feet tested
  For each prosthetic foot, patients will fill out a questionnaire, which is a modified form of the standardized prosthesis evaluation questionnaire (PEQ). The PEQ is a clinically-validated, self-report questionnaire used to assess the prosthesis and life with the prosthesis.
  Questions are evaluated on a Likert scale (ie, "Strongly disagree" to "Strongly agree") which will be converted to numerical values. A low score represents a poor rating (the patient did not like the device) and a high score represents a strong rating.
  The overall outcome measure is the difference in total score (totaled across all questions) between each foot condition. The score for an individual foot represents an overall evaluation of that prosthesis, which we will average across participants and compare between feet. The difference in scores evaluates the feasibility of the prototype foot compared with the subject's own, daily-use prosthesis as well as the commercially available control prosthetic foot.

CONTACTS AND LOCATIONS:
Overall Officials: Amos G Winter, PhD, Principal Investigator — Massachusetts Institute of Technology
Locations (1):
- Hanger Clinic, Salt Lake City, Utah, United States

IPD SHARING:
Plan to Share IPD: No
The aggregated data will be kept for several years in order to compare the performance of this prototype with the performance of future prototypes. Data collected will be subjective feedback, information about prosthetic foot alignment, and biomechanical data about walking patterns, none of which is particularly sensitive.
  While participant data is not particularly sensitive, it pertains to intellectual property of new prosthetic foot designs, and we will not be making the individual participant data (IPD) available to other researchers.

REFERENCES:
- See also: Page with overview of the MIT researcher's project — https://www.gear.mit.edu/prosthetic-foot